CLINICAL TRIAL: NCT03725618
Title: Immunogenicity of Fractional One-fifth and One-half Doses of Yellow Fever Vaccine Compared to Full Dose in Children 9-23 Months Old
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Infectious Disease Institute, Kampala, Uganda (Other); MRC/UVRI and LSHTM Uganda Research Unit (Other); Ministry of Health, Uganda (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017-197
Record Dates: First submitted 2018-10-12; First posted 2018-10-31 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Yellow Fever
MeSH Terms: conditions — Yellow Fever

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- One-fifth fractional dose (Experimental): One-fifth fractional dose (0.1 ml) of Yellow Fever 17DD Vaccine administered subcutaneously
  Interventions: Biological: Yellow Fever 17DD Vaccine
- One-half fractional dose (Experimental): One-half fractional dose (0.25 ml) of Yellow Fever 17DD Vaccine administered subcutaneously
  Interventions: Biological: Yellow Fever 17DD Vaccine
- Full dose (Experimental): Full dose (0.5 ml) of Yellow Fever 17DD Vaccine administered subcutaneously
  Interventions: Biological: Yellow Fever 17DD Vaccine

INTERVENTIONS:
Biological: Yellow Fever 17DD Vaccine — live attenuated vaccine based on the 17DD strain

SUMMARY:
A randomized clinical trial comparing fractional dose Yellow Fever vaccination to the full dose among children aged 9-23 months in Uganda. Children will have immune response assessed at baseline, 4 weeks, and 12 months after vaccination.

Enrolled participants will be randomized to one of three arms:

A. One-fifth fractional dose (0.1 ml) administered subcutaneously B. One-half fractional dose (0.25 ml) administered subcutaneously C. Full dose (0.5 ml) administered subcutaneously

DETAILED DESCRIPTION:
Yellow fever (YF) is a potentially fatal disease causing some 29,000 - 60,000 deaths in Africa alone in 2013. Vaccination with the YF vaccine is the most effective way of preventing YF and a single full dose of vaccine provides life-long protection. Indeed, over half a billion doses of the YF vaccine have been successfully used worldwide since its introduction over 80 years ago in the 1930s, including in children <2 years of age. The World Health Organization (WHO) recommends that YF vaccine be administered to all people ≥ 9 months of age. It should be noted that four YF vaccines are prequalified for use by WHO. Between 2007 and 2016, more than 105 million people have been vaccinated against YF in 14 African countries, including millions of children 9-24 months of age. Each year 6 million doses of YF vaccine are placed into an emergency stockpile to assist in the rapid response and control of outbreaks. During 2016, large outbreaks of YF in Angola and the Democratic Republic of Congo (DRC) depleted the stockpile multiple times and led to critical shortages in YF vaccine. Given the acute vaccine shortage, the World Health Organization (WHO) reviewed available data and determined that the use of fractional dose YF vaccination was a safe and effective option for mass vaccination to control outbreaks. Fractional 1/5th dose of YF vaccine manufactured by BioManguinhos, 17DD, was then used in a campaign targeting 8 million people in DRC's capital city of Kinshasa. However, only persons aged 2 years of age and older were given the fractional dose as there were no data regarding its use in children. To optimize vaccination coverage and vaccine use in outbreak responses, studies of fractional dose YF vaccine effectiveness in children less than 2 years of age were assessed as a research priority by the Strategic Advisory Group of Experts on Immunization (SAGE).

To address this critical information need, the investigators will conduct a randomized clinical trial comparing fractional dose 17DD YF vaccination to the full dose among children aged 9-23 months in Uganda. Exclusion criteria will include children who have previously received YF vaccine or who have contraindications or precautions to YF vaccination.

Enrolled participants will be randomized to one of three arms:

A. One-fifth fractional dose (0.1 ml) administered subcutaneously B. One-half fractional dose (0.25 ml) administered subcutaneously C. Full dose (0.5 ml) administered subcutaneously

The one-fifth and one-half doses of YF vaccine were both recommended for further research by WHO and YF vaccine experts.

Three large public health centers that provide vaccination through the Ministry of Health of Uganda's Expanded Programme on Immunization will be selected in Kampala and nearby districts as study sites. Blood samples (3 ml) will be collected from participants before vaccine administration as well as at follow-up visits 4 weeks and 12 months after vaccination. Presence of YF virus-specific neutralizing antibodies in the collected specimens will be determined using the plaque reduction neutralization test (PRNT). Seroconversion will be defined as seronegative participants (<1:10 titers) at enrollment who become seropositive (≥1:10) at 4 week follow-up. An immune response will be defined as either participants that seroconvert or participants who demonstrate a four-fold or greater change in titers between the baseline and 4 week specimens, e.g. a change from 1:20 to 1:80. The proportion of children seroconverting in each of the fractional dose arms will be compared to the full dose arm using a non-inferiority test. The safety profile also will be described for both solicited and unsolicited adverse events following immunization (AEFIs).

The investigators will collect data on all illnesses encountered by study participants during the first 28 days post-vaccination to assess potential AEFI as recommended by the WHO. Since almost all AEFI occur during the first 2 weeks post-vaccination, parents/guardians will be interviewed at 2 weeks to determine if there are any signs and symptoms that could be consistent with a serious AEFI known to be associated with YF vaccination. In addition, parents will be asked to take their child's temperature twice during the day and complete a structured diary card to document all of their child's signs and symptoms for pre-specified and un-specified adverse events during the first 2 weeks. This will be reviewed by study staff at the 2 week visit as described above. At the 4 week visit, parents/guardians will be asked about illnesses during the interval between their 2 week and 4 week visits as described above. In addition, parents will be reminded and instructed at all interactions during the first 28 days after vaccination to call study staff anytime on the 72-hour study phone line and bring their child directly to the study hospital if they develop any condition(s) requiring medical attention during the first 28 days after vaccination. Any adverse events observed will be reported to the national reporting system.

ELIGIBILITY:
Inclusion Criteria:

1. Age 9 to 23 months at the time of enrollment
2. Intent to stay in the health center catchment area and availability to do study visits at 2 weeks, 4 weeks, and 12 months after enrollment date
3. Informed consent signed by parent/guardian for child's participation in the study, including blood sample collections at 4 week and 12 month visits post-vaccination
4. Willingness of parent/guardian to be contacted by study personnel by telephone and through home visits if they cannot be reached by telephone.

Exclusion Criteria:

1. Verbal or written report of previous vaccination against YF
2. Verbal or documented history of YF disease
3. Contraindication for YF vaccine including:

   1. Allergy to eggs, gelatin, or neomycin
   2. Severe immune deficiency immunological including symptomatic HIV infection and HIV- infected persons with CD4 T-cell counts ≤200 cells/ mm³, primary immunodeficiencies, having received immunosuppressive doses of oral or injectable corticosteroids (or equivalent), having received immunomodulatory or chemotherapeutic agents
   3. Thymus disorder
   4. History of malignant neoplasm or recent hematopoietic stem cell transplantation
   5. Serious illness/fever (mild illness without fever is not an exclusion criterion)
4. Administration of immunoglobulins or other blood derivative within 6 months of enrollment in the study or during the study

   a. Exception: children with a history of Kawasaki disease who received gammaglobulin cannot be enrolled if they received it in the previous 11 months.
5. Administration of any other attenuated viral vaccine in the month prior to enrollment, or if the administration of any other attenuated viral vaccine is expected during the month after enrollment. Note: the administration of measles vaccine on the same day as YF vaccination is not a contraindication; however, if Uganda introduces measles-rubella vaccine (MR), participants will not be able to receive MR on the same day as YF vaccine due to possible interference between rubella and YF vaccine. In this situation, children will have to delay study enrollment until 1 month after MR vaccination.
6. Participating in another clinical drug trial of a drug, vaccine, or medical device
7. Severely underweight defined as ≤ 3rd percentile in the height/weight tables
8. Severe reaction to prior vaccination
9. Any chronic or other condition that, in the opinion of the study staff, represents a health risk to the participant or interferes with the evaluation of the response to the vaccine

   -

Ages: 9 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1788 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Immune response at 4 weeks in terms of seroconversion following vaccination | 4 weeks post vaccination
  Assess whether seroconversion following one-fifth (0.1 ml) and one-half (0.25 ml) doses of YF 17DD vaccine is non-inferior to seroconversion following a full dose (0.5 ml) at 4 weeks post-vaccination in children aged 9 - 23 months. Study endpoints at 4 weeks will be the following: Seroconversion will be defined as seronegative participants (plaque reduction neutralization test with a 50% cut-off (PRNT50) < 10) at enrollment who become seropositive (PRNT50 ≥ 10) at 4 week follow-up. A boosted response will be defined as baseline-positive participants who demonstrate a four-fold or greater change in YF virus-specific titers between the baseline and 4 week specimens, e.g. a change from 1:20 to 1:80.

SECONDARY OUTCOMES:
Immune response at 12 months in terms of seroconversion following vaccination | 12 months post vaccination
  Assess whether the proportion of baseline seronegative children that are seropositive following one-fifth (0.1 ml) and one-half (0.25 ml) doses of YF 17DD vaccine is non-inferior to the proportion seropositive following a full dose (0.5 ml) of vaccine at 12 months post-vaccination. At 12 months, the endpoint will be a plaque reduction neutralization test with a 50% cut-off ( PRNT50) ≥ 10 as evidence of seropositivity

OTHER OUTCOMES:
Titers at 4weeks and 12 months | 4 weeks and 12 months
  • Compare the geometric mean antibody titers following the fractional doses to the geometric mean titer following the full dose at 4 weeks and 12 months post vaccination
Frequency of adverse events following vaccination | 1 hour, 3 days, 14 days, 28 days
  Compare frequency of adverse events for pre-defined conditions associated with yellow fever vaccine and serious adverse events associated following vaccination, as defined by Brighton Criteria and WHO guidelines, in the trial between the 3 study arms

CONTACTS AND LOCATIONS:
Locations (1):
- Centers for Disease Control and Prevention, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Casey RM, Harris JB, Ahuka-Mundeke S, Dixon MG, Kizito GM, Nsele PM, Umutesi G, Laven J, Kosoy O, Paluku G, Gueye AS, Hyde TB, Ewetola R, Sheria GKM, Muyembe-Tamfum JJ, Staples JE. Immunogenicity of Fractional-Dose Vaccine during a Yellow Fever Outbreak - Final Report. N Engl J Med. 2019 Aug 1;381(5):444-454. doi: 10.1056/NEJMoa1710430. Epub 2018 Feb 14. PMID 29443626
- [Derived] Lee SE, Najjengo M, Shaum A, Sekiziyivu AB, Carlock G, Casey RM, Lubega I, Tumwine C, Twinomuhwezi-Oyet E, Nakato WN, Sciarratta CN, Hyde TB, Chu SY, Doshi RH, Kambugu A, Gidudu JF. Adverse events following immunization (AEFI) with fractional one-fifth and one-half doses of yellow fever vaccine compared to standard dose in children 9-23 months old in Uganda, 2019-2022 - final report. Vaccine. 2026 Feb 27;74:128131. doi: 10.1016/j.vaccine.2025.128131. Epub 2026 Jan 8. PMID 41512502